CLINICAL TRIAL: NCT07066839
Title: Pharmacokinetics and Bioavailability of Three Chrysin Formulations in Healthy Adults
Brief Title: Chrysin Bioavailability and Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isura (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-11-002CR
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Bioavailability and Pharmacokinetics; Safety After Oral Intake
Keywords: chrysin; pharmacokinetics; bioavailability; micellar delivery; natural health products; caco-2 permeability; safety; dietary supplements

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to interventions in a crossover design to assess the pharmacokinetics over 24 hours; subsequently, the safety of LipoMicel Chrysin intervention with the higher bioavailability is evaluated in a subsequent single-arm, 30-day trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LipoMicel Chrysin (Experimental): Each participant receives their treatment i.e., LipoMicel Chrysin at a total dose of 1000 mg chrysin. Treatments are consumed with a glass of water (approx. 200mL), followed by a standardized breakfast (diet-controlled condition) 2 hours post-dose. Capillary whole blood samples are collected at different time points up to 24 hours post-dose. A washout period of at least 7 days between each treatment is used.
  Interventions: Dietary Supplement: LipoMicel Chrysin
- Non-micellar Chrysin (Experimental): Each participant receives their treatment i.e., Non-Micellar Chrysin at a total dose of 1000 mg chrysin. Treatments are consumed with a glass of water (approx. 200mL), followed by a standardized breakfast (diet-controlled condition) 2 hours post-dose. Capillary whole blood samples are collected at different time points up to 24 hours post-dose. A washout period of at least 7 days between each treatment is used.
  Interventions: Dietary Supplement: Non-Micellar Chrysin
- Standard Unformulated Chrysin (Experimental): Each participant receives their treatment i.e., Standard Unformulated Chrysin at a total dose of 1000 mg chrysin. Treatments are consumed with a glass of water (approx. 200mL), followed by a standardized breakfast (diet-controlled condition) 2 hours post-dose. Capillary whole blood samples are collected at different time points up to 24 hours post-dose. A washout period of at least 7 days between each treatment is used.
  Interventions: Dietary Supplement: Standard/Unformulated Chrysin

INTERVENTIONS:
Dietary Supplement: LipoMicel Chrysin — A maximum single oral dose of 1000 mg chrysin
  Arms: LipoMicel Chrysin
Dietary Supplement: Non-Micellar Chrysin — A maximum single oral dose of 1000 mg chrysin
  Arms: Non-micellar Chrysin
Dietary Supplement: Standard/Unformulated Chrysin — A maximum single oral dose of 1000 mg chrysin
  Arms: Standard Unformulated Chrysin

SUMMARY:
This study seeks to evaluate and compare the pharmacokinetics of a micellar chrysin formulation (LipoMicel Chrysin) with that of a non-micellar chrysin formulation as well as a standard/unformulated chrysin supplement. The study also seeks to determine the short-term effects and safety of daily oral supplementation of LipoMicel Chrysin in healthy adult volunteers over a 30-day study period.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged 21-65 years
* healthy, good physical condition
* voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

* use of anti-inflammatory or non-steroidal anti-inflammatory drugs
* previous history of cardiovascular disease or acute or chronic inflammatory disease
* use of antioxidant or polyphenol supplements or cholesterol-lowering agents
* change of diet habits or lifestyle (diet, physical activity, etc.)
* alcohol or substance abuse history
* use of nicotine or tobacco
* participation in another investigational study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Cmax: maximum plasma concentration | 0 (baseline; pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 24 hours (post-dose)]
  To determine the gastrointestinal absorption of orally ingested chrysin in healthy adult volunteers and compare the peak plasma concentration (Cmax) with that of other capsules containing chrysin.
AUC: the area under the concentration-time curve | 0 (baseline; pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 24 hours (post-dose)]
  To determine the gastrointestinal absorption of orally ingested chrysin in healthy adult volunteers and compare the Area under the plasma concentration versus time curve (AUC) with that of other capsules containing chrysin.
Tmax: the time point of maximum plasma concentration | 0 (baseline; pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 24 hours (post-dose)]
  To determine the gastrointestinal absorption of orally ingested chrysin in healthy adult volunteers and compare the time point of maximum plasma concentration (Tmax)

SECONDARY OUTCOMES:
Alanine aminotransferase (ALT) | [Time Frame: 0 (baseline; pre-dose), week 1, week 2, week 3 and week 4 (post-dose)]
  To evaluate changes in liver function based on ALT.
Aspartate aminotransferase (AST) | [Time Frame: 0 (baseline; pre-dose), week 1, week 2, week 3 and week 4 (post-dose)]
  To evaluate changes in liver function based on AST.
Total bilirubin (TB) | [Time Frame: 0 (baseline; pre-dose), week 1, week 2, week 3 and week 4 (post-dose)]
  To evaluate changes in liver function based on total bilirubin.
Serum creatinine | [Time Frame: 0 (baseline; pre-dose), week 1, week 2, week 3 and week 4 (post-dose)]
  To evaluate changes in kidney function based on serum creatinine.
Glomerular filtration rate (GFR) | [Time Frame: 0 (baseline; pre-dose), week 1, week 2, week 3 and week 4 (post-dose)]
  To evaluate changes in kidney function based on GFR.
Fasting blood glucose | [Time Frame: 0 (baseline; pre-dose), week 1, week 2, week 3 and week 4 (post-dose)]
  To evaluate changes in blood glucose levels based on fasting blood glucose.
HbA1c | [Time Frame: 0 (baseline; pre-dose), week 1, week 2, week 3 and week 4 (post-dose)]
  To evaluate changes in blood glucose levels based on HbA1c.
Total cholesterol | [Time Frame: 0 (baseline; pre-dose), week 1, week 2, week 3, and week 4 (post-dose)]
  To evaluate changes in lipid profile based on total cholesterol.
Triglycerides | [Time Frame: 0 (baseline; pre-dose), week 1, week 2, week 3, and week 4 (post-dose)]
  To evaluate changes in lipid profile based on triglycerides.
Low-density lipoprotein (LDL) cholesterol | [Time Frame: 0 (baseline; pre-dose), week 1, week 2, week 3, and week 4 (post-dose)]
  To evaluate changes in lipid profile based on LDL.
High-density lipoprotein (HDL) cholesterol | [Time Frame: 0 (baseline; pre-dose), week 1, week 2, week 3, and week 4 (post-dose)]
  To evaluate changes in lipid profile based on HDL.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Solnier, PhD, Principal Investigator — Isura
Locations (1):
- ISURA, Burnaby, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No